CLINICAL TRIAL: NCT06141993
Title: Clinical Validation of a Circulating Tumor Cell AR Therapy Resistance Assay in Men With Metastatic Castration Resistant Prostate Cancer (ARCTIC)
Brief Title: ARCTIC: Liquid Biomarkers in the Prospective Androgen Receptor Signaling Inhibitors (ARSI) Resistance Clinical Trials
Acronym: ARCTIC
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Wisconsin, Madison (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00111532
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Cancer Metastatic; Castration-resistant Prostate Cancer
Keywords: Circulating Tumor Cells (CTC); Androgen-receptor signaling inhibitors (ARSI); Metastatic castration resistant prostate cancer (mCRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Men with progressive metastatic castration resistant prostate cancer (mCRPC): Men with progressive metastatic castration resistant prostate cancer (mCRPC) and starting standard of care therapy with a second androgen receptor (AR) inhibitor (typically enzalutamide or abiraterone acetate) will have blood collected for circulating tumor cell (CTC) assessments and other research assessments at baseline, 12 weeks and upon disease progression.

SUMMARY:
This study will follow men with metastatic castration resistant prostate cancer throughout their standard of care treatment for their disease to determine if the presence of different genes or proteins can predict which patients respond to the cancer treatment they receive. As tumors grow and begin to spread, they may release cells into patients' bloodstream. These cells are called "circulating tumor cells", or CTCs. CTCs can be used to look for differences in "biomarkers" (genes or proteins that may change based on how a person is or is not responding to treatment). The purpose of this research study is to learn whether scientists can use biomarkers from CTCs to predict which tumors will respond to certain hormonal therapies. Participants will have blood collected and provide an archival sample from a previous tumor biopsy. The researchers will compare biomarkers from participants who responded well to treatment to those who responded poorly in order to answer the research question.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in this study only if all of the following criteria apply:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Patients with pure small cell/neuroendocrine tumors of the prostate are not permitted.
2. Radiographic evidence of metastatic disease by CT, MRI, or PET imaging.
3. Prior documented disease progression on one potent AR inhibitor (darolutamide, abiraterone, enzalutamide, or apalutamide or combinations of these) in any disease setting (mHSPC, nmCRPC, mCRPC) based on sequential PSA rises or radiographic progression.
4. Planned therapy with either standard of care enzalutamide and/or abiraterone acetate or another potent AR inhibitor (darolutamide, apalutamide if available) within the coming 6 weeks
5. Castrate levels of testosterone (<50 ng/dl) at most recent assessment and/or documented ongoing Androgen Deprivation Therapy.
6. Evidence of disease progression based on a rising PSA on or following most recent therapy as evidenced by the following:

   1. Consecutive PSA rises at least 2 weeks apart
   2. Minimum PSA of 1.0 ng/dl prior to entry
7. Age > 18 years.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of intercurrent or past medical or psychiatric illness including active stage IV malignancy that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Unwillingness to be followed longitudinally for serial CTC biomarker studies.
3. Life expectancy < 6 months
4. Planned combination therapy with radiation or other systemic therapies other than ADT and bone health agents.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes men with progressive metastatic castration resistant prostate cancer (mCRPC) as defined in the eligibility criteria listed below. Participants will enroll at one of three locations: Duke University, University of Wisconsin Madison and Memorial Sloan Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of progression-free survival (PFS) between biomarker positive and negative participants | Through completion of participant participation, up to 3 years
  PFS which is defined as the time from date of study enrollment to radiographic or clinical progression or death. Radiographic progression will be defined by Prostate Cancer Working Group 3 (PCWG3) criteria for soft tissue and bone metastases and will not include PSA changes alone. Clinical progression will be defined as clinical deterioration requiring a change in therapy, such as a pathologic fracture or symptomatic skeletal event or pain progression in the absence of imaging progression.

SECONDARY OUTCOMES:
Comparison of overall survival between biomarker positive and negative participants | Through completion of participant participation, up to 3 years
  Overall survival is defined as time from date of study enrollment to date of death or last contact.
Comparison of the proportion of participants that achieve a >50% PSA declines from baseline between biomarker positive and negative participants | Through completion of participant participation, up to 3 years
  PSA decline will be assessed per PCWG3
Comparison of soft tissue response between biomarker positive and negative participants | Through completion of participant participation, up to 3 years
  Soft tissue response will be assessed per RECIST 1.1.
Comparison of duration of therapy between biomarker positive and negative participants | Through discontinuation of current therapy, up to 3 years
  Time from initiation to discontinuation of therapy
Number of emergent molecular lesions in CTCs that consistently emerge during subsequent AR therapy progression in men with mCRPC | At disease progression, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No